CLINICAL TRIAL: NCT03692494
Title: The Effects of Adding Expiratory Muscle Strength Training in Voice Therapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI did decided reorganize the methodology for this study and will resubmit in the future.
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Adam Lloyd, Speech Pathologist, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20171103
Record Dates: First submitted 2018-09-26; First posted 2018-10-02 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-02

CONDITIONS: Dysphonia; Unilateral Vocal Cord Paralysis
MeSH Terms: conditions — Dysphonia; Vocal Cord Paralysis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Unilateral vocal fold paralysis standard of care voice therapy (Experimental): The participants will receive the standard of voice therapy including improved breath coordination, sustained humming and vowels, vocal glides, resonant voice therapy, and relations techniques.
  Interventions: Other: Standard of care voice therapy
- Unilateral paralysis standard of care voice therapy plus EMST (Experimental): The participants will receive the standard of voice therapy including improved breath coordination, sustained humming and vowels, vocal glides, resonant voice therapy, and relations techniques. EMST consists of blowing into respiratory device at a measure threshold pressure. As strength improves threshold resistance will be increased.
  Interventions: Other: Standard of care voice therapy; Other: Expiratory muscle strength training (EMST)
- Parkinson's disease standard of care voice therapy plus EMST (Experimental): The participants will receive the standard of voice therapy including improved breath coordination, sustained humming and vowels, vocal glides, resonant voice therapy, and relations techniques. EMST consists of blowing into respiratory device at a measure threshold pressure. As strength improves threshold resistance will be increased.
  Interventions: Other: Standard of care voice therapy; Other: Expiratory muscle strength training (EMST)

INTERVENTIONS:
Other: Standard of care voice therapy — Exercises will include improved breath coordination, sustained humming and vowels, vocal glides, resonant voice therapy, and relaxation techniques to the neck and shoulder
Other: Expiratory muscle strength training (EMST) — EMST150 used at 75% of their maximum expiratory pressure. Participants will be directed to perform 5 sets of 5 breaths, 5 days per week, for 5 weeks, at the pressure threshold established in therapy. Maximum expiratory pressure will then be determined at the beginning of each therapy session and recalibration of the device will be performed if indicated.
  Arms: Parkinson's disease standard of care voice therapy plus EMST; Unilateral paralysis standard of care voice therapy plus EMST

SUMMARY:
Evaluate if adding expiratory muscle strength training to traditional voice therapy for individuals with dysphonia due to glottal insufficiency improves maximal expiratory pressure, acoustic and aerodynamic measures (i.e. amplitude, maximum phonation time, peak expiratory flow), and voice related quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with glottic insufficiency.
* Adequate cognition evidenced by score of 24 or higher on the Mini-Mental State Examination (MMSE) survey to determine if the subject has the mental capacity to participate in therapy
* Completed voice combination evaluation with speech pathologists and otolaryngologist.
* Individuals 18 years of age or older

Exclusion Criteria:

* Adults unable to consent
* Non English or Spanish speakers
* Pregnant women
* Prisoners
* Individuals with significant uncontrolled chronic and progressive respiratory diseases including COPD, interstitial lung disease, and cystic fibrosis.
* Individuals with uncontrolled blood pressure.
* Individuals with significant GI disease and/or gastroesophageal surgery with the exception of well-controlled GERD.
* Individuals with a history of abdominal hernia.
* Individuals with difficulty complying due to neuropsychological dysfunction (e.g., severe depression, psychosis).
* Individuals with other neurological disorders and/or neuromuscular disease other than Parkinson's Disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Maximum expiratory pressure | 16 weeks
  Maximum expiratory pressure, in cm of H2O, will be measured to evaluate how much pressure a participant can blow into a respiratory pressure meter.
Amplitude | 16 weeks
  Amplitude of voice, in decibels, will be measured using Voice Range Profile on Kay Pentax CSL and will be compared to gender matched normative values for normal and loud volumes.

SECONDARY OUTCOMES:
Fundamental frequency | 16 weeks
  Fundamental frequency, measured in herz, will be obtained using the Analysis of Dysphonia in Speech and Voice on Kay Pentax Computerized Speech Lab.
Dynamic pitch range | 16 weeks
  Dynamic pitch range will be measured using Voice Range Profile on Kay Pentax Computerized Speech Lab.
Cepstral Peak Prominence (CPP) | 16 weeks
  Cepstral Peak Prominence will be obtained using the Analysis of Dysphonia in Speech and Voice on Kay Pentax Computerized Speech Lab.
Cepstral spectral index of dysphonia (CSID) | 16 weeks
  Cepstral spectral index of dysphonia, will be obtained using the Analysis of Dysphonia in Speech and Voice on Kay Pentax Computerized Speech Lab.
Voice Handicap Index | 16 weeks
  This is quality of life assessment tool quantifying perception of the impact of their vocal disorder on various aspects of lifestyle. It is 30-questions in length and is divided into 3 subscales including emotional, physical, and functional, divided into 10 questions each. Each question scored from 0-4. Total score range from 0-120. Higher score indicates increased handicap.
Maximum phonation time | 16 weeks
  The patient will be asked to inhale deeply and sustain the vowel /a/ at a comfortable loudness level for a many seconds as possible.
Peak expiratory flow rate | 16 weeks
  Peak expiratory flow rate, measured in units of liters per minute, will be measured for purposes of measuring cough function.

CONTACTS AND LOCATIONS:
Overall Officials: Adam T Lloyd, SLP-D, MM, MA, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No